CLINICAL TRIAL: NCT03836521
Title: The International Multicenter Bicuspid Aortic Valve Stenosis Transcatheter Aortic Valve Replacement Registry
Brief Title: Bicuspid Aortic Valve Stenosis Transcatheter Aortic Valve Replacement Registry
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Raj Makkar, Profssor of Medicine, University of California, Cedars-Sinai Medical Center
Other Study IDs: Pro00047203
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Bicuspid Aortic Valve
MeSH Terms: conditions — Bicuspid Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Transcatheter aortic valve replacement

SUMMARY:
The objective of this study is to evaluate the procedural and clinical outcomes of patients with bicuspid aortic valve stenosis undergoing transcatheter aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years.
2. Severe aortic stenosis with bicuspid anatomy.
3. NYHA≥2 and/or syncope and/or angina.
4. Patient judged by the Heart Team as indicated for TAVR.

Exclusion Criteria:

1. Age <18 years
2. Asymptomatic patients
3. Pure aortic regurgitation.

Ages: 19 Years to 129 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients presenting with severe and symptomatic bicuspid aortic valve stenosis or mixed disease
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-08-15 (Actual); Primary Completion 2028-08-15 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
Death | 1 month
  Death from any cause
Death | 1 year
  Death from any cause
Death | 2 years
  Death from any cause
Death | 3 years
  Death from any cause
Death | 4 years
  Death from any cause
Death | 5 years
  Death from any cause

SECONDARY OUTCOMES:
Death from cardiac cause | 1 month
  Death from cardiac cause
Death from cardiac cause | 1 year
  Death from cardiac cause
Death from cardiac cause | 2 years
  Death from cardiac cause
Death from cardiac cause | 3 years
  Death from cardiac cause
Death from cardiac cause | 4 years
  Death from cardiac cause
Death from cardiac cause | 5 years
  Death from cardiac cause
Stroke | 1 month
  disabling and non-disabling stroke
Stroke | 1 year
  disabling and non-disabling stroke
Stroke | 2 years
  disabling and non-disabling stroke
Stroke | 3 years
  disabling and non-disabling stroke
Stroke | 4 years
  disabling and non-disabling stroke
Stroke | 5 years
  disabling and non-disabling stroke
Repeat hospitalization | 1 month
  Number of hospitalizations
Repeat hospitalization | 1 year
  Number of hospitalizations
Repeat hospitalization | 2 years
  Number of hospitalizations
Repeat hospitalization | 3 years
  Number of hospitalizations
Repeat hospitalization | 4 years
  Number of hospitalizations
Repeat hospitalization | 5 years
  Number of hospitalizations
Bleeding | 1 month
  Life-threatening or major bleeding rate
Bleeding | 1 year
  Life-threatening or major bleeding rate
Bleeding | 2 years
  Life-threatening or major bleeding rate
Bleeding | 3 years
  Life-threatening or major bleeding rate
Bleeding | 4 years
  Life-threatening or major bleeding rate
Bleeding | 5 years
  Life-threatening or major bleeding rate
Vascular complication | 1 month
  Major vascular complication
Vascular complication | 1 year
  Major vascular complication
Vascular complication | 2 years
  Major vascular complication
Vascular complication | 3 years
  Major vascular complication
Vascular complication | 4 years
  Major vascular complication
Vascular complication | 5 years
  Major vascular complication
Acute kidney injury (stage 2 or 3) | 1 month
Acute kidney injury (stage 2 or 3) | 1 year
Acute kidney injury (stage 2 or 3) | 2 years
Acute kidney injury (stage 2 or 3) | 3 years
Acute kidney injury (stage 2 or 3) | 4 years
Acute kidney injury (stage 2 or 3) | 5 years
Prosthetic regurgitation by Doppler echocardiography | at discharge
Prosthetic regurgitation by Doppler echocardiography | 1 month
Prosthetic regurgitation by Doppler echocardiography | 1 year
Prosthetic regurgitation by Doppler echocardiography | 2 years
Prosthetic regurgitation by Doppler echocardiography | 3 years
Prosthetic regurgitation by Doppler echocardiography | 4 years
Prosthetic regurgitation by Doppler echocardiography | 5 years
Mean aortic valve gradient by Doppler echocardiography | 1 month
Mean aortic valve gradient by Doppler echocardiography | 1 year
Mean aortic valve gradient by Doppler echocardiography | 2 years
Mean aortic valve gradient by Doppler echocardiography | 3 years
Mean aortic valve gradient by Doppler echocardiography | 4 years
Mean aortic valve gradient by Doppler echocardiography | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Yoon SH, Kim WK, Dhoble A, Milhorini Pio S, Babaliaros V, Jilaihawi H, Pilgrim T, De Backer O, Bleiziffer S, Vincent F, Shmidt T, Butter C, Kamioka N, Eschenbach L, Renker M, Asami M, Lazkani M, Fujita B, Birs A, Barbanti M, Pershad A, Landes U, Oldemeyer B, Kitamura M, Oakley L, Ochiai T, Chakravarty T, Nakamura M, Ruile P, Deuschl F, Berman D, Modine T, Ensminger S, Kornowski R, Lange R, McCabe JM, Williams MR, Whisenant B, Delgado V, Windecker S, Van Belle E, Sondergaard L, Chevalier B, Mack M, Bax JJ, Leon MB, Makkar RR; Bicuspid Aortic Valve Stenosis Transcatheter Aortic Valve Replacement Registry Investigators. Bicuspid Aortic Valve Morphology and Outcomes After Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2020 Sep 1;76(9):1018-1030. doi: 10.1016/j.jacc.2020.07.005. PMID 32854836